CLINICAL TRIAL: NCT05839613
Title: How Personalized Medicine Based on Pharmacogenetics and Therapeutic Drug Monitoring Can Reduce Relapse Rate in Patients WITH schizophreniA: An Analytical, Experimental, Prospective, Comparative, Adaptive Randomized, Open-label, Multicenter Clinical Trial
Brief Title: PhaRmacOgenetics and Therapeutic Drug Monitoring In SchizophrEnia
Acronym: PROMISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A01015-38
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Patients With Schizophrenia
MeSH Terms: interventions — Drug Monitoring

STUDY DESIGN:
Intervention Model Description: The design of this study is a two parallel arms, followed during 12 months, randomized (1:1 ratio) as follow:
  * 200 patients in the experimental group with PG/TDM intervention (PG/TDM group).
  * 200 patients in Control group with the SOC group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PG/TDM group (Experimental): experimental group with PG/TDM analysis results avalaible
  Interventions: Diagnostic Test: Therapeutic Drug Monitoring (TDM) and Pharmacogenetics (PG)
- blinded group (Experimental): experimental group with PG/TDM analysis results blinded
  Interventions: Diagnostic Test: Therapeutic Drug Monitoring (TDM) and Pharmacogenetics (PG)

INTERVENTIONS:
Diagnostic Test: Therapeutic Drug Monitoring (TDM) and Pharmacogenetics (PG) — Pharmacogenetics (PG) is the study of genetic differences in drug met-abolic pathways Therapeutic Drug Monitoring (TDM) is the quantification and interpre-tation of drug concentration in blood to optimize pharmacotherapy

SUMMARY:
Schizophrenia is a severe chronic mental disorder with a long-term treatment. Most antipsychotic (AP) drugs are effective for only 30% to 60% of patients and for many drugs, treatment selection remains a "trial-and-error" process.The main result of treatment inefficiency is relapse, the recurrence of acute symptoms after a period of partial or complete remission.

Pharmacogenetics (PG) is the study of genetic differences in drug met-abolic pathways which can affect individual responses to drugs, both in terms of therapeutic effect as well as adverse effects. PG testing could therefore identify patients at potentially high risk of relapse allowing the opportunity of an individualized prescription. In this study, PG was shown to improve the safety profile of AP treatments in patients presenting PM or UM CYP variants, by reducing associated side effects. Therapeutic Drug Monitoring (TDM) is the quantification and interpretation of drug concentration in blood to optimize pharmacotherapy . For drugs with established therapeutic reference ranges (TRR) or with a narrow therapeutic index, it makes sense to measure drug concentrations in blood for dose titration after initial prescription or after dose change. Non adherence is a recurrent problem in the management of schizophrenia, leading to reduced quality of life and increased risk of relapse. TDM is recognized as a direct reliable measure for drug adherence and can be an additional support after a therapy adjustment. Additionally, TDM can be useful to educate patients and make them more aware of their treatment. Finally, TDM is likely to ensure a better tolerance and fewer side effects for APs, while allowing a better efficacy. However, evidence on the clinical impact of this tool in schizophrenic population is lacking and randomized clinical trials are needed to confirm it.

Finally, relapses occur frequently in schizophrenia and the cost for a relapsing schizophrenic patient is estimate over 4 times higher than for a non-relapsing patient, highlighting the importance of cost-effective care strategies.

When separately used PG testing or TDM alone, might not be sufficient to ensure the clinical utility and cost-effectiveness of these tests. We hypothesize that individualized medicine including the association of PG testing with TDM (PG/TDM intervention), on the most commonly prescribed AP drugs, can reduce relapse rate at one year while being cost-effective.

DETAILED DESCRIPTION:
The variability of treatment response for both efficacy and side effects is multifactorial. Non-pharmacological aspects, such as psychological and social implications, influence drug response but at the pharmacological level, drug response results from the interaction of genetic (e.g. drug-metabolizing enzymes, drug transporters, drug targets), personal (e.g. age, sex, disease states, treatment adherence) and environmental factors (e.g. smoking, diet, alcohol habits, drug-drug interactions) that produce interindividual differences in term of pharmacokinetics and pharmacodynamics (de Leon 2009). Moreover, non-adherence is linked to the pathology itself and also to adverse drug reactions. Because the development of new APs is slow, it is of paramount importance to use the currently available drugs as effectively as possible. An important aspect of effective use is dose personalization because, owing to interindividual differences in drug metabolism, the dose required to achieve optimal concentration of APs varies substantially between patients (Jukic et al., 2019). Two main tools are available for the optimization of APs exposure: PG testing and TDM.

PG testing can help reduce the uncertainty inherent in psychiatric pharmacotherapy by detecting genetic factors that predict clinical response and side effects, such as genetic variations that impact drug-metabolizing enzymes, drug transporters or drug targets (Evans et Johnson 2001; Evans et Relling 1999). PG is the study of genetic differences in drug metabolic pathways which can affect individual responses to drugs, both in terms of therapeutic effect as well as adverse effects (Nebert 1999). In France, PG is now well implanted in university hospitals and anti-cancer institutions as well as in certain private medical laboratories (Picard et al. 2017). According to the medical and scientific report of the Biomedecine Agency (ABM), 56 laboratories reported PG activity in 2019 compared with 47 laboratories with such activity in 2015 and 38,091 patients were tested in 2019 (vs 18,777 in 2015) (Annual activity report of postnatal genetic, ABM, 2019). Interpretation requires expertise in genetics and in pharmacology. Depending on the degree of enzymatic deficiency, treatment can be reduced from onset, or an alternative drug can be proposed if the deficiency is severe. The therapeutic attitude will be modulated depending on the clinical context (disease gravity, existence or not of a therapeutic alternative).

The identification of robust clinical criteria and biomarkers (e.g., genetic variants) for guiding treatment choice has been the objective of a number of research efforts and part of the resulting findings were recently incorporated in guidelines. In a recent review, author's aims to provide an overview of the available studies focused on the genetic predictors of antidepressants response, the current clinical applications of antidepressants PG and possible future developments (Zanardi et al. 2020). The future clinical approach in psychiatry as well as in other fields of medicine is indeed represented by precision medicine, that aims to integrate genetic, environmental, clinical and lifestyle individual factors in order to personalize treatments.

Cytochromes P450 2D6 and 2C19 genetic polymorphisms are well-known to influence APs pharmacokinetics (Crettol et al. 2014). CYP2D6 and CYP2C19 haplotypes are assigned a star-allele (*) nomenclature to allow for the standardization of genetic polymorphism annotation (Robarge et al. 2007). Then, diplotype, which is the summary of inherited maternal and paternal star-alleles, allows to categorized CYP2D6 and CYP2C19 into functional groups based on the predicted activity of the encoded enzyme (Hicks et al. 2017, 2015). The predicted phenotype is influenced by the expected function of each reported allele in the diplotype, making it possible to differentiate four groups of phenotypes: extensive metabolizer (EM), who have classically two functional alleles; intermediate metabolizer (IM), with classically one inactive allele and one causing a reduced rate of metabolism; poor metabolizer (PM), carrying two inactive alleles with no functional activity and ultrarapid metabolizer (UM), who have classically an increased enzymatic function (Bondy et Spellmann 2007). To date, the interest of identification of PM and UM is recently growing and should help to individualize therapeutic regimens and current guidelines of the CPIC and DPWG require dose adjustment according to CYP2D6, CYP2C19 or CYP3A4/3A5 genetic variants (www.pharmGKB.org). Based on the currently available information, Arranz, Salazar et Hernández (2021) has presented that PG intervention should be reduced to APs' dose adjustment according to the genetically predicted metabolic status (CYPs' profile) of the patient. Growing evidence suggests that such interventions will reduce APs' side-effects and increase treatment safety. Despite this evidence, the use of PG in psychiatric wards is minimal. Hopefully, further evidence on the clinical and economic benefits, the development of clinical protocols based on PG information, and improved and cheaper genetic testing will increase the implementation of PG guided prescription in clinical settings.

Two recent randomized clinical trial failed to demonstrate the impact of PG alone on clinical improvement in schizophrenic patients. Jürgens et al. (2019) described a randomized clinical trial witch the aim was to assess whether routine genetic testing for CYP2D6 and CYP2C19 (CYP testing) improves AP drug treatment in patients with schizophrenia in terms of improved drug persistence, a surrogate for tolerability and effectiveness, compared with clinically guided treatment. The authors concluded that routine CYP2D6 and CYP2C19 genotyping had no effect on AP drug persistence. In the study of Arranz et al. (2019), no evidence of greater efficacy of PG intervention was observed. However, results show that PG may improve the safety profile of AP treatments in patients presenting PM or UM CYP variants, by reducing associated side effects. The PG intervention described in this study may be particularly useful when considering treatment with APs with one major metabolic pathway, and therefore more susceptible to be affected by functional variants of CYP metabolizing enzymes. These recent studies confirm the fact that PG alone can only partially explain the variability pharmacokinetic of APs.

TDM has a long standing history in clinical psychiatry and has been proved to be a reasonably adequate tool for the management of individual variability in psychotropic drug response (Albers et Ozdemir 2004; Hiemke et al. 2018). Non-response at therapeutic doses, uncertain drug adherence, suboptimal tolerability, or pharmacokinetic drug-drug interactions are typical indications for TDM (Hiemke et al. 2018). Additionally, TDM can be useful to educate patients and make them more aware of their treatment. Finally, TDM is likely to ensure a better tolerance and fewer side effects for antipsychotics drugs, while allowing a better efficacy.

For drugs with established TRR or with a narrow therapeutic index, it makes sense to measure drug concentrations in blood for dose titration after initial prescription or after dose change. Even without a specific problem, there is sufficient evidence that TDM has beneficial effects for patients treated with the following drugs: lithium, tricyclic antidepressants, several APs or anticonvulsants (Hiemke et al. 2018; de Leon, Armstrong, et Cozza 2006). Indeed, since more than a decade, the TDM task force of the working group on neuropsychopharmacology (Arbeitsgemeinschaft fuer Neuropsychopharmakologie und Pharmakopsychiatrie, AGNP) has worked out consensus guidelines to assist psychiatrists and laboratories involved in psychotropic drug analysis to optimise the use of TDM of psychotropic drugs and recommendations for genotyping (Baumann et al. 2004; Hiemke et al. 2018, Schoretsanitis et al. 2020). Five research-based levels of recommendation were defined with regard to routine monitoring of plasma concentrations for dose titration of 65 psychoactive drugs: (1) strongly recommended, (2) recommended, (3) useful, (4) probably useful and (5) not recommended (Baumann et al. 2004). A list of recommended TRR was also established (table 4 of the guideline). AP strongly recommended (1) and recommended (2) are: amisulpride, aripiprazole, bromperidol (not available in France), chlorpromazine, clozapine, flupentixol, fluphenazine, haloperidol, olanzapine, paliperidone, perazine (not available in France), perphenazine (not available in France), quetiapine, risperidone, sertindole (not available in France since 2007), sulpiride and ziprasidone (not available in France).

To conclude, measuring drug concentrations in blood is advantageous compared to other methods, since it tells the prescribing psychiatrist whether the drug is in the body at a concentration that is potentially sufficient to provide the expected clinical response, i.e. pharmacodynamics effect. However, evidence on the clinical impact of this tool in schizophrenic population is lacking and randomized clinical trials are needed to confirm it.

Taking together, PG and TDM display marked synergy in the following areas of medical therapeutics (Albers et Ozdemir 2004; Ozdemir, Shear, et Kalow 2001):

* To explain the mechanism of pharmacodynamic variability related to drug targets;
* To provide pharmacokinetic exposure beyond the study sample in various populations, including evaluations in population extreme metabolizers (i.e. UM and PM);
* To explain and predict drug distribution to tissues outside the plasma compartment by genetic testing of drug transporters;
* To provide drug exposure prior to drug administration and make appropriate dose adjustments early in the course of pharmacotherapy, thereby reducing the time-lag for therapeutic response and avoiding acute drug toxicity that may occur after several doses of atypical APs;
* To provide the risk for inhibitory and inductive drug/drug or drug/food interaction potential by genetic testing and elucidation of the drug metabolism pathways that contribute to APs disposition in vivo.

The most important indications for combining CYP450 genotyping and TDM are presented by Zanardi et al. (2020): 1) when prescribing a drug with a narrow therapeutic index and high risk of toxicity; 2) when a drug has wide interindividual variability in metabolism and a considerable risk of toxicity; 3) a post hoc genotyping when the patient presents unusual plasma concentrations of the drug or its metabolite(s), indicating a possible alternation of drug metabolism or the lack of adherence to the prescribed dose (so-called pseudo-resistance); the latter should of course be checked before CYP450 genotyping.

Therefore on APs area, on the one hand, PG biomarkers, included in prescribing guidelines, could represented an important step towards precision psychiatry. On the other hand, TDM, important and cost-effective tool (Hiemke et al. 2018), should be integrated with genetic testing and clinical evaluation in order to adjust dose and optimize pharmacotherapy.

PG testing or TDM alone, might not be sufficient to ensure the clinical utility and cost-effectiveness of these tests, when separately used in patients suffering from schizophrenia.

Combined PG and TDM testing should improve acute and long-term treatment, prediction of therapeutic response, possible correlations with treatment outcome, reduction of side effects, and monitoring of treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤ 60 years.
2. Diagnostic of schizophrenia according to DSM-5.
3. The clinical situation of the patient justifies a modification of his AP treatment according to the judgment of the attending psychiatrist (relapsing patients or patients in maintenance phase judged clinically stable by the attending psychiatrist but not optimally treated e.g. non- satisfactory treatment regarding symptoms or adverse events (AEs), Gaebel et al. 2010) or non-compliant patient or patient who has stopped the AP treatment.
4. The patient is to receive a prescription for at least one of the following molecules in oral or injectable forms: aripiprazole, olanzapine, paliperidone, quetiapine, risperidone, amisulpride
5. Women and men of reproductive potential must agree to use highly effective contraception during the study.

Exclusion Criteria:

1. Patients who do not meet the schizophrenia criteria as defined in the DSM-5.
2. Patient with current prescription of clozapine.
3. Patient who are in maintenance phase and optimally treated e.g. satisfactory treat- ment regarding symptoms or AEs (Gaebel et al. 2010).
4. Previous PG testing used for drug therapy adjustment.
5. Pregnant or breastfeeding woman.
6. Subject refusing to give written informed consent.
7. Adults protected by the law
8. Subject non-affiliated to the French health insurance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Clinical worsening | 12 months
  Clinical worsening as defined by CGI-S score ≥ 5 and an increase of 25 % from base- line in the total score of the PANSS or an increase of 10 points if the baseline score was 40 or less Csernansky criteria (Csernansky et al. 2002)
Hospitalization | 12 months
  Hospitalization due to worsening of psychotic symptoms
Risk of suicide | 12 months
  Risk of suicide as defined by a CGI-SS score ≥ 6 (much worse)
Violent behavior | 12 months
  Violent behavior resulting in clinically significant self-injury, injury to another person, or property damage
Serious Adverse Events | 12 months
  APs related Serious Adverse Events (SAE)

SECONDARY OUTCOMES:
Number of relapses | 12 months
  Total number of relapses on accounting criteria: number of hospitalization, number of suicide attempts and number of violent behavior
Time to relapse | 12 months
  Time to relapse: time (days) until first relapse
Remission rate | 12 months
  • Remission rate from Andreasen and adapted by Bo (Andreasen et al. 2005; Bo et al. 2017) defined as the achievement of a score of 3 (mild), 2 (minimal), or 1 (absent) for eight items on the PANSS: P1, P2, P3, N1, N4, N6, G5 and G9 RSWG criteria
Therapeutic range | 12 months
  Rate of results of drug concentration in the TRR
Clinical change | 12 months
  Change from baseline of PANSS total score > to 25 % (Leucht et al. 2005)
Genetic polymorphism | 12 months
  Description: exploratory study of polymorphisms of genes and transporters (ABCB1, COMT, DRD2, HTR...) involved in the pharmacokinetics or pharmacodynamics of the APs